CLINICAL TRIAL: NCT04450823
Title: From Short-term Surgical Missions Towards Sustainable Partnerships. A Survey Among Members of Foreign Teams
Brief Title: From Short-term Surgical Missions Towards Sustainable Partnerships
Status: Completed | Type: Observational
Sponsor: Global Surgery Amsterdam (Other)
Responsible Party: Principal Investigator, Matthijs Botman, Principal investigator, Global Surgery Amsterdam
Other Study IDs: 2020-01
Record Dates: First submitted 2020-06-20; First posted 2020-06-30 (Actual); Results first posted 2020-08-05 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-11

CONDITIONS: Global Surgery; Medical Missions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention study, survey amongst health workers

SUMMARY:
Introduction: Recently, the devastating consequences of neglected surgical care in global health became apparent with an estimated five billion people lacking access to safe surgical and anesthesia care. Traditionally, short-term surgical missions were the predominant strategy how surgical care was supported in Low- and Middle-Income Countries. Although surgical missions have been criticized in recent literature they are still being performed on a large scale. The aim of this study is to provide recommendations for persons and organizations involved in surgical mission on how to strengthen surgical care in LMICs in the future.

Method: An online survey was developed for members of foreign teams. Data was collected on 5 topics, consisting of: 1) basic characteristics of the missions, 2) main activities, 2) follow-up and reporting, 3) the local registration process for foreign teams and 4) collaboration with local stakeholders.

ELIGIBILITY:
Inclusion Criteria:

Members of foreign teams, that did participate in at least one short-term surgical mission in a hospital in a LMIC

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: An international group of members of foreign teams, that did participate in at least one short-term surgical mission in a hospital in a LMIC
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Global surgery amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared anonymously on this platform as requested by the journal of submission (int,. journal of surgery)
Supporting Information: Study Protocol
Time Frame: ASAP

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was June through October of 2019
Groups:
- Experts: Included were English speaking experienced members of foreign teams and local team members from LMIC, that did participate in at least one short-term surgical mission in a hospital in a LMIC.
Period: Overall Study
Arm/Group | Experts
Started | 61
Completed | 58
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- All Participants of the Study: Included were English speaking experienced members of foreign teams and local team members from LMIC, that did participate in at least one short-term surgical mission in a hospital in a LMIC.
Arm/Group | All Participants of the Study
Number analyzed (Participants) | 58
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43 [32 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 38
Race (NIH/OMB) [Count of Participants; unit: Participants] — We did not register Race as a variable in this study
  Participants
    American Indian or Alaska Native | NA — not considered to be relevant in this study
    Asian | NA — not considered to be relevant in this study
    Native Hawaiian or Other Pacific Islander | NA — not considered to be relevant in this study
    Black or African American | NA — not considered to be relevant in this study
    White | NA — not considered to be relevant in this study
    More than one race | NA — not considered to be relevant in this study
    Unknown or Not Reported | NA — not considered to be relevant in this study
Nationality [Count of Participants; unit: Participants] — in the survey provided answer on the question what is your nationality:
  Participants
    Dutch | 33
    German | 5
    British | 4
    American | 4
    Australian | 2
    South African | 2
    Tanzanian | 1
    Lebanese | 1
    Nigerian | 1
    Danish | 1
    Indian | 1
    Haitian | 1
    Ethiopian | 2
Profession [Count of Participants; unit: Participants]
  plastic surgeons | 23
  orthopedic surgeons | 9
  general surgeons | 4
  local doctors/surgeons in training | 12
  anaesthetists | 5
  nurses | 2
  physiotherapists | 2
  NGO executive officer | 1
Number of missions performed [Mean (Full Range); unit: missions] — by the respondent provided number of surgical missions performed in the past by the respondent him- or herself
  missions | 6 [3 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Q7: Country Where the Last Mission Took Place
Description: Answer on the question: What was the country where your last mission took place?
Time Frame: approximately 20 minutes
Measure: Count of Participants; unit: Participants
Groups:
- All Included Participants of the Study: Included were English speaking experienced members of foreign teams and local team members from LMIC, that did participate in at least one short-term surgical mission in a hospital in a LMIC.
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 58
Participants
  Burkino fase | 2
  Bangladesh | 2
  Cambodia | 1
  Ecuador | 1
  Ethiopia | 3
  Gaza | 1
  Guinea | 9
  Guinee Bissau | 2
  Haiti | 1
  Indonesia | 2
  Laos | 1
  Lebanon | 1
  Malawi | 1
  Morocco | 2
  Nigeria | 3
  Peru | 1
  Rwanda | 1
  Senegal | 2
  Sierra Leone | 3
  Sri LAnka | 1
  Tanzania | 13
  Uganda | 4
  Vietnam | 1

2. Primary Outcome: Q8: Name of the Place and Hospital Where the Last Mission Took Place
Description: List with names of the places and hospitals where the last mission took place
Time Frame: approximately 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 58
Participants
  Paul VI, Ouaga | 1
  Sekou Toure Regional Referral hospital | 1
  Harapan, pematang Siantar, Sumatera Bissau Hospita | 1
  Haydom Lutheran Hospital, Haydom | 9
  St Josephs, Kitgum | 1
  Comprehensive Health Centre, totoro Abeokuta. | 1
  Sengerema hospital, sengerema | 3
  Masanga Hospital | 3
  Pius VI, Ouagadougou | 1
  St Francis hospital Mutolere | 1
  Pemantang siantar, rumah sakit harapan | 1
  Virgen de la puerta | 1
  Gatagara | 1
  Rach Gia | 1
  Yekatit 12 hospital, Addis Ababa | 1
  Guercif, Morocco; | 1
  Munshiganj, Bangladesh | 1
  Ambroseli Hospital Kalongo | 2
  Conakry, Port. Mercy Ships | 1
  Mahossot Hospiatl Vientiane | 1
  Vavuniya General Hospital | 1
  Guayaquil | 1
  Bekhazi Medical Center, Beirut | 1
  Bissau teaching hospital | 1
  Conakry | 5
  Malamulo Hospital | 1
  Dhaka Medical College Hospital, Dhaka | 1
  Yekatit 12 | 1
  CSC, Phnom Penh | 1
  Africa Mercy | 1
  Mercships | 1
  Hopital National Donka, Conakry | 1
  Africa Mercy, Conakry | 1
  Exeter | 1
  Mangu Hospital, Mangu Plateau state | 1
  Cocin, Mangu | 1
  University Hospital Basel, Switzerland | 1
  Yekatit 12 Hospital, Addis Ababa | 1
  Shifa Hospital, Gaza City | 1
  MSF burn hospital in Port-au-Prince, Haiti | 1

3. Primary Outcome: Q9: Number of Participants Per Organization
Description: Name of the organization that supported the last mission of the participant
Time Frame: approximately 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 58
Participants
  Bridge the Gap Foundation | 1
  B-first | 1
  Doctors of the World | 11
  Global Smile Foundation | 3
  Harapan Jaya | 2
  Ka Dounia Dia | 2
  MAP | 1
  Mercy Ships | 12
  Mission Restore | 1
  MSF | 1
  Njokuti | 3
  Operation Hernia | 1
  Orthopaedic Outreach | 1
  Pan-African Academy of Christian Surgeons | 1
  Project Harar | 2
  Resurge | 1
  Interplast Holland | 6
  Simba Health | 2
  Stichting 'Op Gelijke Voet' | 1
  Trinitas Health Care Partners | 1
  Mission without a supporting NGO | 4

4. Primary Outcome: Q10: Countries Where the NGOs Are Based
Description: List of countries where the supporting NGOs of the last mission are based
Time Frame: approximately 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 58
Participants
  Netherlands | 29
  USA | 17
  No supporting NGO | 4
  UK | 4
  Australia | 1
  France | 1
  Nigeria | 1
  Sierra Leone | 1

5. Primary Outcome: Q11: Importance of Potential Activities
Description: Points provided (1-4) for four potential activities of a visiting team (more points = more important activity) The points provided by all participants are summed per specific activity and the total scores are compared
  The four potential activities are:
  * Treat patients yourself
  * Provide surgical equipment and consumables for the local team
  * Provide free treatment
  * Facilitate teaching of local staff
  Scale with importance of potential activities. Maximum score: 4x58 = 232
Time Frame: approximately 20 minutes
Measure: Number; unit: score on a scale
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 58
score on a scale
  Treat patients yourself | 157
  Provide surgical equipment and consumables for the | 153
  Provide free treatment | 175
  Facilitate teaching of local staff | 210

6. Primary Outcome: Q12: Activities That Where Missing in Question 11.
Description: Respondents that were missing this activity as an option in question 11
  Total number of respondents that were missing an activity: 29
  Activities that were missing:
  * Financial collaboration
  * Advocacy
  * Academic collaboration
  * Sustainability
  * Collaboration with local staff
  * Follow-up
Time Frame: approximately 20 minutes
Population: Question 12 was asked to all participants but only 29 stated that an activity was missing in question 11
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 29
Participants
  Financial collaboration | 1
  Advocacy | 2
  Academic collaboration | 4
  Sustainability | 5
  Collaboration with local staff | 8
  Follow up | 9

7. Primary Outcome: Q13. Medical Registration is Required in the Host Country
Description: Medical registration in the host country is required for specialists performing short-term reconstructive missions
  Participants of the survey were asked what they think of this statement:
  * Strongly agree
  * Agree
  * Neither agree nor disagree
  * Disagree
  * Strongly disagree
Time Frame: approximately 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 58
Participants
  Strongly agree | 28
  Agree | 16
  Neither agree nor disagree | 7
  Disagree | 7
  Strongly disagree | 0

8. Primary Outcome: Q14: The Process of Obtaining Medical Registration Was Straightforward
Description: The Process of Obtaining Medical Registration Was Straightforward
  Participants of the survey were asked what they think of this statement:
  * Strongly agree
  * Agree
  * Neither agree nor disagree
  * Disagree
  * Strongly disagree
Time Frame: approximately 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 58
Participants
  Strongly agree | 8
  Agree | 19
  Neither agree nor disagree | 16
  Disagree | 10
  Strongly disagree | 5

9. Primary Outcome: Q15: Collaboration
Description: What can you say about the collaboration between authorities in LMICs and visiting surgical teams?
  Participants of the survey were asked to choose one of the following answers on this question:
  * collaboration is present but improvement is needed
  * there is no collaboration and it should be developed as a priority
  * collaboration has no benefits nor disadvantages
  * collaboration will likely be more harmful than beneficial for the mission
Time Frame: approximately 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 58
Participants
  collaboration is present but improvement is neede | 39
  there is no collaboration and it should be develop | 16
  collaboration has no benefits nor disadvantages | 3
  -collaboration has no benefits nor disadvantages | 1

10. Primary Outcome: Q16. What Should Have a Higher Priority in the Hospital of Your Last Mission?
Description: What should have a higher priority in the hospital of your last mission ?
  Respondents were asked to choose on the these two answers:
  Teaching in anesthesia care or teaching in surgical care
Time Frame: approximately 20 minutes
Population: 5 respondents did't make a choice In the comments section 9 respondents declared that preferable both should be equally addressed
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 53
Participants
  Surgical care | 31
  Anaesthesia care | 22

11. Primary Outcome: Q17. A Structured Follow-up Strategy is Required
Description: A structured follow-up strategy (>6 months) of patients is required for short-term reconstructive surgical missions.
  Participants of the survey were asked what they think of this statement:
  * Strongly agree
  * Agree
  * Neither agree nor disagree
  * Disagree
  * Strongly disagree
Time Frame: approximately 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 58
Participants
  Strongly agree | 37
  Agree | 17
  Neither agree nor disagree | 4
  Disagree | 0
  Strongly disagree | 0

12. Primary Outcome: Q18. One Month After the Mission, an Official Report is Recommended
Description: One month after the mission, an official report on the outcome including all complications encountered is recommended for all missions.
  Participants of the survey were asked what they think of this statement:
  * Strongly agree
  * Agree
  * Neither agree nor disagree
  * Disagree
  * Strongly disagree
Time Frame: approximately 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 58
Participants
  Strongly agree | 39
  Agree | 16
  Neither agree nor disagree | 2
  Disagree | 1
  Strongly disagree | 0

13. Primary Outcome: Q19. A Written Long-term Strategy is Recommended at the Start of a New Project.
Description: A written long-term strategy (>5 years) with clear goals, developed by the visiting team and the local actors together, is recommended at the start of a new project.
  Participants of the survey were asked what they think of this statement:
  * Strongly agree
  * Agree
  * Neither agree nor disagree
  * Disagree
  * Strongly disagree
Time Frame: approximately 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 58
Participants
  Strongly agree | 37
  Agree | 17
  Neither agree nor disagree | 4
  Disagree | 0
  Strongly disagree | 0

14. Primary Outcome: Q20. Suggestions to Improve the Impact of Short Term Reconstructive Missions.
Description: What would you suggest to improve the impact of short term reconstructive missions?
  The answers were categorized and the three most mentioned categories are:
  * Teaching of local staff
  * Follow-up
  * Building sustainable partnerships
  The three activities were mentioned in total 68 times in the comments The distribution among the three categories is shown below
Time Frame: approximately 20 minutes
Population: the 58 participants mentioned the top three activities 68 times
Measure: Number; unit: answers mentioning this activity
Arm/Group | All Included Participants of the Study
Number analyzed (Participants) | 58
answers mentioning this activity
  Teaching of local staff | 24
  Follow-up | 10
  Building sustainable partnerships | 34

ADVERSE EVENTS:
Time Frame: 5 months
Description: Adverse Events data was not collected.
  Because this study is a survey, there is no intervention group
Arm/Group | Experts
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
An important limitation of this study is that most of the respondents are medical doctors from HICs.

Another possible 'selection bias' that could have occurred concerns (over-) representation of experts from the Netherlands.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT04450823/Prot_000.pdf